CLINICAL TRIAL: NCT02172131
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Doses of 0.5 μg, 2.5 μg, 5 μg, 10 μg, 15 μg, 20 μg, 25 μg and 30 μg BI 1744 CL (Calculated as Free Base) Given as Intravenous Infusion Over 30 Minutes to Healthy Male Subjects. A Single-centre, Single-blind, Placebo-controlled, Randomised Study.
Brief Title: Safety, Tolerability and Pharmacokinetics Study of BI 1744 CL in Healthy Male Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1222.7
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
MeSH Terms: interventions — olodaterol

ARMS (2):
- BI 1744 CL (Experimental): Single rising dose of BI 1744 CL as intravenous (i.v.) infusion
  Interventions: Drug: BI 1744 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1744 CL
  Arms: BI 1744 CL
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate safety, tolerability, and pharmacokinetics (PK) of single i.v. doses of BI 1744 CL

ELIGIBILITY:
Inclusion Criteria:

* Healthy male based upon a complete medical history, including the physical examination, regarding vital signs (blood pressure (BP), pulse rate (PR)), 12-lead ECG measurement, and clinical laboratory tests. There is no finding deviating from normal and of clinical relevance. There is no evidence of a clinically relevant concomitant disease.
* Age ≥21 and ≤45 years
* BMI ≥18.5 and <30 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR, and ECG measurements) deviating from normal and of clinical relevance
* Evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to the drug or its excipients) as judged clinically relevant by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least 1 month or less than 10 half-lives of the respective drug prior to medication
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to medication
* Participation in another trial with an investigational drug within 2 months prior to medication
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days as judged by the investigator
* Alcohol abuse (more than 40 g alcohol a day)
* Drug abuse
* Blood donation (more than 100 mL blood within 4 weeks prior to medication or during the trial)
* Excessive physical activities within 1 week prior to randomisation or during the trial
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of the study centre.

The following exclusion criteria are specific for this study due to the known class side effect profile of ß2-mimetics:

* Asthma or history of pulmonary hyperreactivity
* Hyperthyrosis
* Allergic rhinitis in need of treatment
* Clinically relevant cardiac arrhythmia
* Paroxysmal tachycardia (>100 beats per minute)

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2006-10; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with abnormal findings in physical examination | Baseline, Day 10 after drug administration
Number of patients with clinically significant changes in vital signs | Baseline and up to day 10 after drug administration
Number of patients with abnormal changes in 12-lead ECG (electrocardiogram) parameters | Baseline and up to day 10 after drug administration
Number of patients with abnormal changes in laboratory parameters | Baseline and up to day 10 after administration
Number of patients with adverse events | Up to day 10
Assessment of tolerability by investigator on a 4-point scale | Day 10 after drug administration

SECONDARY OUTCOMES:
AUC (area under the concentration-time curve of the analyte in plasma at different time points) | Up to 48 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) | Up to 48 hours after drug administration
tmax (time from dosing to maximum measured concentration) | Up to 48 hours after drug administration
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | Up to 48 hours after drug administration
λz (terminal rate constant in plasma) | Up to 48 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | Up to 48 hours after drug administration
MRT (mean residence time of the analyte in the body after intravenous administration) | Up to 48 hours after drug administration
CL (total clearance of the analyte in plasma after intravascular administration) | Up to 48 hours after drug administration
V (apparent volume of distribution at different time points following an intravascular dose) | Up to 48 hours after drug administration
Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) | Up to 96 hours after drug administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | Up to 96 hours after drug administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | Up to 96 hours after drug administration